CLINICAL TRIAL: NCT03848754
Title: Pracinostat in Combination With Gemtuzumab Ozogamicin (PraGO) in Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Brief Title: Pracinostat and Gemtuzumab Ozogamicin (PraGO) in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sameem M. Abedin, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO 33922
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Relapsed Adult AML
Keywords: acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab; SB939 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pracinostat 45 mg with Gemtuzumab Ozogamicin (Experimental): * Gemtuzumab Ozogamicin Induction: GO 3 mg/m^2 on Day 1, 4, and 7
  * Pracinostat Induction: 45 mg administered orally 3 days a week with 48 hours between dosing for 3 consecutive weeks, followed by 1 week of rest, in 28-day cycles. We will utilize a 3+3 design to determine the safe dose of pracinostat in combination with fixed dose GO. If there are no DLTs in the first three patients, the dose of pracinostat will be escalated to 60mg. Escalation to the next dose level will be done only after the third patient on the previous dose level has been observed for 28 days, and no DLTs were noticed. If there is 1 DLT, an additional 3 patients will be tested at same dose level. If there are ≥ 2 DLTs in 3 or 6 patients, the study will be placed on hold. If there is < 2 DLTs in the first 3 or 6 patients, the dose of pracinostat will be escalated to 60mg. If there are no DLTs in the first 3 patients at 60 mg, an additional 3 patients will be enrolled to ensure 6 patients are treated at the MTD.
  Interventions: Drug: Gemtuzumab Ozogamicin 3 mg/m^2; Drug: Pracinostat - 45 mg
- Pracinostat 60 mg with Gemtuzumab Ozogamicin (Experimental): * Gemtuzumab Ozogamicin Induction: GO 3 mg/m^2 on Day 1, 4, and 7
  * Pracinostat: 60 mg administered orally 3 days a week with 48 hours between dosing for 3 consecutive weeks, followed by 1 week of rest, in 28-day cycles.
  We will utilize a 3+3 design to determine the safe dose of pracinostat in combination with fixed dose GO. If there are no DLTs in the first three patients, the dose of pracinostat will be escalated to 60mg. Escalation to the next dose level will be done only after the third patient on the previous dose level has been observed for 28 days, and no DLTs were noticed. If there is 1 DLT, an additional 3 patients will be tested at same dose level. If there are ≥ 2 DLTs in 3 or 6 patients, the study will be placed on hold. If there is < 2 DLTs in the first 3 or 6 patients, the dose of pracinostat will be escalated to 60mg. If there are no DLTs in the first 3 patients at 60 mg, an additional 3 patients will be enrolled to ensure 6 patients are treated at the MTD.
  Interventions: Drug: Gemtuzumab Ozogamicin 3 mg/m^2; Drug: Pracinostat - 60 mg
- Gemtuzumab Ozogamicin Monotherapy Maintenance (Experimental): Response will be assessed through bone marrow biopsy on Day 28. Patients achieving at least a partial remission marrow will be offered up to 5 cycles of maintenance therapy. Maintenance should begin no later than 42 days after initial induction.
  **Gemtuzumab Ozogamicin Maintenance: 2 mg/m^2 intravenous administration on day 1, in a 28-day cycle.
  Interventions: Drug: Gemtuzumab Ozogamicin 2 mg/m^2
- Pracinostat with Gemtuzumab Ozogamicin Maintenance (Experimental): Response will be assessed through bone marrow biopsy on Day 28. Patients achieving at least a partial remission marrow will be offered up to 5 cycles of maintenance therapy. Maintenance should begin no later than 42 days after initial induction.
  * Gemtuzumab Ozogamicin Maintenance: 2 mg/m^2 intravenous administration on day 1, in a 28-day cycle.
  * Pracinostat Maintenance: (In addition to GO, only if induction dose escalation occurs) 45 mg orally 3 days a week with 48 hours between dosing, for three consecutive weeks, followed by 1 week of rest, in a 28-day cycle.
  Interventions: Drug: Gemtuzumab Ozogamicin 2 mg/m^2; Drug: Pracinostat - 45 mg

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin 3 mg/m^2 — GO 3 mg/m^2 on Day 1, 4, and 7
  Maintenance: 2mg/m2 intravenous administration on day 1, in a 28-day cycle.
  Other Names: Mylotarg
  Arms: Pracinostat 45 mg with Gemtuzumab Ozogamicin; Pracinostat 60 mg with Gemtuzumab Ozogamicin
Drug: Gemtuzumab Ozogamicin 2 mg/m^2 — GO 2 mg/m^2 on Day 1 of a 28-day cycle.
  Other Names: Mylotarg
  Arms: Gemtuzumab Ozogamicin Monotherapy Maintenance; Pracinostat with Gemtuzumab Ozogamicin Maintenance
Drug: Pracinostat - 45 mg — Induction: 45mg administered orally 3 days a week with 48 hours between dosing (e.g., Monday, Wednesday, and Friday) for three consecutive weeks, followed by 1 week of rest, in 28-day cycles.
  Arms: Pracinostat 45 mg with Gemtuzumab Ozogamicin; Pracinostat with Gemtuzumab Ozogamicin Maintenance
Drug: Pracinostat - 60 mg — Escalation: 60 mg administered orally three days a week with 48 hours between dosing (e.g., Monday, Wednesday, and Friday) for three consecutive weeks, followed by one week of rest, in 28-day cycles.
  Arms: Pracinostat 60 mg with Gemtuzumab Ozogamicin

SUMMARY:
This is a prospective, single-center phase 1 clinical study aimed at determining the maximum-tolerated dose and safety of the combination of gemtuzumab ozogamicin (GO) and pracinostat (P) in patients with relapsed/refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
Relapsed/Refractory AML (RR-AML) is a serious medical condition where overall less than 10% survive beyond five years. Among RR-AML patients ineligible for intensive chemotherapy, this problem is magnified, and survival is measured in months. Hence, there is an urgent need for more efficacious and tolerable therapies for RR-AML.

The majority of AML expresses the cluster of differentiation 33 (CD33) surface antigen. Gemtuzumab Ozogamicin (GO) is a recombinant, humanized anti-CD33 monoclonal antibody covalently attached to the cytotoxic antitumor antibiotic calicheamicin. GO binds to the CD33 antigen on AML cells forming a complex which is internalized, resulting in the intracellular delivery of calicheamicin. Calicheamicin then binds to DNA in the minor groove, inciting DNA double strand breaks and triggering cell death. GO was recently FDA approved for patients with AML who cannot tolerate intensive chemotherapy, and additionally received FDA approval in the RR-AML setting on the basis of a modest complete response (CR) rate of 26% [95% confidence interval (CI) 16-40%].

The investigators are studying whether the addition of the Histone deacetylase (HDAC) inhibitor pracinostat to GO is safe, and effective. HDACs plays important role in transcription regulation and in the pathogenesis of cancer. HDAC inhibitors induces histone hyperacetylation, resulting in an open chromatin structure and restore transcription of critically silenced genes. In AML, early clinical trials using single agent Pracinostat have demonstrated potential activity against the disease.

In the context of GO, the investigators hypothesize HDAC inhibition may potentially synergize with GO to improve response against AML. Through HDAC inhibition mediated histone unwinding, open chromatin could allow for increased DNA delivery of calicheamicin within AML blasts and increased apoptosis. Further, pre-clinical data suggests HDAC inhibition could also increase CD33 expression in myeloid leukemia cells, thereby allowing for increased GO binding to AML blasts. This is the basis for the combination of these agents.

ELIGIBILITY:
Inclusion Criteria:

1. Morphologically documented AML or secondary AML [from prior conditions such as myelodysplastic syndrome (MDS), myeloproliferative neoplasm (MPN)] or therapy related AML (t-AML), as defined by World Health Organization (WHO) criteria.
2. Age ≥60 years, with relapsed/refractory AML to at least one line of therapy. Patients with antecedent MDS who progressed to AML while on hypomethylating agent therapy will also be eligible.
3. Age 18-59 years with relapsed/refractory AML to at least two lines of intensive induction chemotherapy, or one line of therapy if deemed unsuitable for further intensive chemotherapy.
4. Patients aged 18 years or older with relapsed AML after allogeneic hematopoietic cell transplantation, if deemed unsuitable for further intensive chemotherapy.
5. Detectable CD33 expression on AML blasts confirmed by flow cytometry.
6. Karnofsky performance status ≥ 60 (or Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) of 2 or less).
7. Adequate organ system function as outlined below:

   * Total bilirubin ≤ 2 x upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN.
   * Serum creatinine ≤ 2 or a serum creatinine clearance ≤ 1.5 x ULN.
   * Baseline EKG with QT-interval corrected (QTcF) ≤ 450ms.
8. Females should be using adequate contraception, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential. Male patient should avoid impregnating a female partner.

   It is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Non-sterilized female patients of reproductive age and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below.

   Female patients must meet one of the following:
   * Postmenopausal for at least one year before the screening visit, or
   * Surgically sterile, or
   * If they are of childbearing potential, agree to practice two effective methods of contraception from the time of signing of the informed consent form through three months after the last dose of study drug, AND
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable contraception methods.)

   Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:
   * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose, OR
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
9. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL).
2. Prior chemotherapy, radiotherapy, or investigative agent within 14 days, or within five half-lives of study entry.

   * Subjects must have recovered from side effects of prior treatment.
   * The use of hydroxyurea for leukoreduction prior to start of dosing is permitted.
3. Hematopoietic Stem Cell Transplantation (HCT) within 60 days of enrollment, or evidence of veno-occlusive disease (VOD) at any time post-transplant, or active graft-versus-host disease requiring systemic immunosuppressive therapy.
4. Life-threatening illness unrelated to AML, or any serious medical or psychiatric illness that could potentially interfere with participation in this study.
5. Active and uncontrolled human immunodeficiency virus (HIV), or chronic Hepatitis B, or Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
The number of subjects experiencing a dose-limiting toxicity. | First 28-day cycle
  Maximum-tolerated (MTD) dose of pracinostat in combination with fixed dose GO induction will be determined by the 3+3 design rules. If there are no dose-limiting toxicities (DLTs) in the first three patients, the dose of pracinostat will be escalated to 60mg. Escalation to the next dose level will be done only after the third patient on the previous dose level has been observed for 28 days, and no DLTs were noticed. If there is 1 DLT, an additional 3 patients will be tested at same dose level. If there are ≥ 2 DLTs in three or six patients, the study will be placed on hold. If there is < 2 DLTs in the first three or six patients, the dose of pracinostat will be escalated to 60mg. If there are no DLTs in the first three patients at 60mg, an additional three patients will be enrolled to ensure six patients are treated at the MTD.

SECONDARY OUTCOMES:
Number of subjects surviving at six months. | 6 Months
  The number of subjects alive at six months.
Number of subjects progression free at 6 months. | 6 Months
  Defined by the IWG.
The number of subjects with a complete response. | Day 28
  A complete response will be defined as bone marrow blasts <5% with absolute neutrophil count ≥1000/L and platelet ≥100,000/mL.
The number of subjects with complete response with incomplete count recovery (CRi). | Day 28
  CRi is defined as CR without platelet recovery or neutrophil recovery. This will be defined as bone marrow blasts <5% with absolute neutrophil count <1000/μL OR platelet <100,000/μL.
The number of subjects with partial remission (PR). | Day 28
  Partial remission (PR) is defined by a decrease of at 50% or more in the percentage of blasts to less than 25% in the bone marrow. and normalized blood counts ( ANC>1000, Platelets>100,000/ml).
The number of subjects with morphologic leukemia-free state (MLFS). | Day 28
  MLFS is bone marrow blasts <5% with absolute neutrophil count <1000/μL AND platelet <100,000/μL.

CONTACTS AND LOCATIONS:
Overall Officials: Sameem Abedin, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No